CLINICAL TRIAL: NCT05409066
Title: A Phase 3, Open-Label Study to Evaluate Safety and Efficacy of Epcoritamab in Combination With Rituximab and Lenalidomide (R2) Compared to R2 in Subjects With Relapsed or Refractory Follicular Lymphoma (EPCORE FL-1)
Brief Title: Study of Subcutaneous Epcoritamab in Combination With Intravenous Rituximab and Oral Lenalidomide (R2) to Assess Adverse Events and Change in Disease Activity in Adult Participants With Follicular Lymphoma
Acronym: EPCORE FL-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-638; 2023-505628-67 (Other: EU CT)
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Follicular Lymphoma (FL)
Keywords: Follicular Lymphoma (FL); Non-Hodgkin's lymphoma (NHL); Lymphoma; Cancer; Epcoritamab; Rituximab; Lenalidomide; EPCORE FL-1; EPCORE
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Epcoritamab Dose A in Combination With R2 (Experimental): Participants will receive epcoritamab Dose A in combination with lenalidomide and rituximab (R2) for 12 cycles (each cycle is 28 days).
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Lenalidomide
- Epcoritamab Dose B in Combination With R2 (Experimental): Participants will receive epcoritamab Dose B in combination with lenalidomide and rituximab (R2) for 12 cycles (each cycle is 28 days). Enrollment is closed for this arm.
  Interventions: Drug: Epcoritamab; Drug: Rituximab; Drug: Lenalidomide
- Lenalidomide and Rituximab (R2) (Active Comparator): Participants will receive lenalidomide and rituximab (R2) for 12 cycles (each cycle is 28 days).
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection
  Arms: Epcoritamab Dose A in Combination With R2; Epcoritamab Dose B in Combination With R2
Drug: Rituximab — Intravenous Infusion
Drug: Lenalidomide — Oral Capsules

SUMMARY:
Follicular Lymphoma (FL) is the second most common B-cell cancer and the most common type of cancer of lymphocytes. Unfortunately, this disease is incurable with conventional treatment and the disease recurs in almost all patients. This study will assess how safe and effective epcoritamab is in combination with lenalidomide and rituximab (R2) in treating adult participants with relapsed or refractory (R/R) FL. Adverse events and change in disease condition will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of FL. Study doctors put the participants in 1 of 3 groups, called treatment arms. Each group receives a different treatment. Enrollment to one of the groups is closed. Around 500 adult participants with R/R FL will be enrolled in approximately 300 sites across the world.

Participants will receive R2 (375 mg/m^2 intravenous infusion of rituximab up to 5 cycles and oral capsules of 20 mg lenalidomide for up to 12 cycles) alone or in combination with subcutaneous injections of epcoritamab for up to 12 cycles (each cycle is 28 days).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score 0 to 2.
* Participant has:

  * Fluorodeoxyglucose-positron emission tomography (FDG-PET) scan demonstrating positive lesion compatible with computed tomography (CT) or magnetic resonance image (MRI)-defined anatomical tumor sites AND
  * >= 1 measurable nodal lesion (long axis > 1.5 cm) or >= 1 measurable extra-nodal lesion (long axis > 1.0 cm) on CT scan or MRI.
* Histologically confirmed classic follicular lymphoma (FL) [previously Grade 1 to 3a FL] stage II, III, or IV with no evidence of histologic transformation to an aggressive lymphoma and CD20+ disease on most recent representative tumor biopsy based on the pathology report.
* Relapsed or refractory (R/R) disease to at least one prior systemic regimen that contained an anti-CD20 monoclonal antibody (mAb) in combination with chemotherapy. (Participant who received only prior anti-CD20 mAb monotherapy and/or radiation therapy is not eligible.)
* Eligible to receive R2 per investigator determination.
* Estimated Creatinine Clearance (CrCl) >= 50 mL/min.

Exclusion Criteria:

* Documented refractoriness to lenalidomide.
* Have lenalidomide exposure within 12 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Best Overall Response (BOR) | Up to approximately 5 years
  BOR is defined as Complete Response (CR) or Partial Response (PR), determined by Lugano criteria, as assessed by an IRC.
Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as duration from the date of randomization to the date of disease progression determined by Lugano criteria by independent review committee (IRC) or death (whichever occurs first).

SECONDARY OUTCOMES:
Percentage of Participants Achieving CR | Up to approximately 5 years
  Percentage of participants who achieve a CR determined per Lugano criteria, as assessed by the IRC prior to the initiation of subsequent anti-lymphoma therapy.
Overall Survival (OS) | Up to approximately 8 years from randomization
  Overall survival is defined as the duration from the date of randomization to the date of the participant's death.
Percentage of Participants Achieving Minimal Residual Disease (MRD) Negativity | Up to approximately 5 years
  MRD negativity rate is defined as the percentage of participants who achieve MRD negative status prior to the initiation of subsequent anti-lymphoma therapy.
Change in Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) | Up to approximately 8 years
  The objective of the FACT-Lym patient-reported outcome (PRO) is to address health-related quality of life issues for adult lymphoma patients. It utilizes a 5-point Like-type scale, with a higher score signifying a higher quality of life.
PFS as Assessed by Investigator | Up to approximately 5 years
  PFS is defined as duration from the date of randomization to the date of disease progression determined by Lugano criteria by investigator or death (whichever occurs first).
Percentage of Participants Achieving BOR as Assessed by Investigator | Up to approximately 5 years
  BOR is defined as CR PR, determined by Lugano criteria, as assessed by an investigator.
Percentage of Participants Achieving CR as Assessed by Investigator | Up to approximately 5 years
  Percentage of participants who achieve a CR determined per Lugano criteria, as assessed by the investigator prior to the initiation of subsequent anti-lymphoma therapy.
Duration of Response (DOR) | Up to approximately 8 years
  DOR is defined as the time from the first occurrence of response (CR or PR) to disease progression or death, whichever occurs first.
Duration of Complete Response (DOCR) | Up to approximately 8 years
  DOR is defined as the time from the first occurrence of CR to disease progression or death, whichever occurs first.
Time to Progression (TTP) | Up to approximately 8 years
  Time to progression is defined as the number of days from the date of study drug start to the date of the first documented disease progression or relapse.
Time to Next Anti-Lymphoma Treatment (TTNLT) | Up to approximately 8 years
  Time to next anti-lymphoma treatment is defined as the number of days from the date of the first documented disease progression or relapse to the date of next anti-lymphoma treatment.
Percentage of Participants Achieving CR at the End of Treatment | Up to approximately 5 years
  Percentage of participants who achieve a CR determined per Lugano criteria, as assessed by the IRC prior to the initiation of subsequent anti-lymphoma therapy.
Time to Response (TTR) | Up to approximately 8 years
  Time to response is defined for participants achieving a CR/PR as the time from starting therapy to first a CR/PR.
Time to Complete Response (TTCR) | Up to approximately 8 years
  Time to complete response is defined for participants achieving a CR/PR as the time from starting therapy to first a CR/PR.
Event-Free Survival (EFS) | Up to approximately 8 years
  EFS is defined as the duration from randomization to disease progression determined by Lugano criteria as assessed by the investigator, initiation of any non-protocol-specified new anti-lymphoma therapy for any reason, or death (whichever occurs first).
Time to next anti-lymphoma treatment (TTNLT) | Up to approximately 8 years
Change in Patient's Global Impression of Severity (PGIS) | Up to approximately 8 years
  PGIS is a self-report measure PGIS reflects a participant's belief about their lymphoma symptoms over the past 7 days. The PGIS is a 5-point scale depicting a participant's rating of overall severity. Participants rate their lymphoma symptoms severity as none, mild, moderate, severe, or very severe.
Change in Patient's Global Impression of Change (PGIC) | Up to approximately 8 years
  PGIS is a self-report measure PGIC reflects a participant's belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement since start of treatment. Participants rate their change as very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Change in EuroQol 5-Dimension Questionnaire, 5-level (EQ-5D-5L) | Up to approximately 8 years
  The EQ-5D-5L descriptive system measures health status and comprises 5 health aspects including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each parameter has 5 response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. This instrument will not be administered during the Survival Follow-Up.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (273):
- United States (31):
  - The University of Arizona Cancer Center - North Campus /ID# 228862, Tucson, Arizona
  - University of Arkansas for Medical Sciences /ID# 227198, Little Rock, Arkansas
  - Alta Bates Summit Medical Center for Research /ID# 229428, Berkeley, California
  - Beverly Hills Cancer Center /ID# 231535, Beverly Hills, California
  - Long Beach Memorial Medical Ct /ID# 228997, Long Beach, California
  - University of Southern California /ID# 227195, Los Angeles, California
  - Valkyrie Clinical Trials /ID# 268502, Los Angeles, California
  - Duplicate_Emory University /ID# 227299, Atlanta, Georgia
  - Hawaii Cancer Care - Waterfront Plaza /ID# 262448, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine /ID# 227248, Chicago, Illinois
  - Goshen Center for Cancer Care /ID# 227189, Goshen, Indiana
  - Community Health Network, Inc. /ID# 259756, Indianapolis, Indiana
  - Our Lady Of The Lake Regional Medical Center /ID# 251393, Baton Rouge, Louisiana
  - University of Maryland, Baltimore /ID# 227191, Baltimore, Maryland
  - Massachusetts General Hospital /ID# 245233, Boston, Massachusetts
  - UMass Memorial Medical Center /ID# 227323, Worcester, Massachusetts
  - Henry Ford Hospital /ID# 227250, Detroit, Michigan
  - St. Luke's Hospital - Chesterfield /ID# 247817, Chesterfield, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 251220, Billings, Montana
  - Morristown Medical Center /ID# 231427, Morristown, New Jersey
  - Roswell Park Cancer Institute /ID# 239128, Buffalo, New York
  - NYU Langone Hospital - Long Island /ID# 253343, Mineola, New York
  - NYU Laura and Isaac Perlmutter Cancer Center /ID# 227322, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 227181, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 227193, New York, New York
  - East Carolina University - Brody School of Medicine /ID# 227192, Greenville, North Carolina
  - University of Oklahoma, Stephenson Cancer Center /ID# 227325, Oklahoma City, Oklahoma
  - Baylor Sammons Cancer Center /ID# 261584, Dallas, Texas
  - Texas Oncology - Northeast Texas /ID# 265890, Tyler, Texas
  - Intermountain Healthcare LDS Hospital /ID# 259948, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 227211, Richmond, Virginia
- Argentina (4):
  - Fundaleu /Id# 229700, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Duplicate_CEMIC /ID# 229697, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 229701, Córdoba, Córdoba Province
  - Clinica de Nefrologia, Urologia y Enfermedades Cardiovasculares /ID# 232124, Santa Fe, Santa Fe Province
- Australia (7):
  - Royal Prince Alfred Hospital /ID# 239272, Camperdown, New South Wales
  - Nepean Hospital /ID# 239093, Kingswood, New South Wales
  - Townsville University Hospital /ID# 231124, Douglas, Queensland
  - Peninsula Private Hospital /ID# 238796, Frankston, Victoria
  - Fiona Stanley Hospital /ID# 231122, Murdoch, Western Australia
  - Royal Perth Hospital /ID# 230456, Perth, Western Australia
  - Hollywood Private Hospital /ID# 251789, Perth, Western Australia
- Austria (3):
  - Universitaetsklinikum St. Poelten /ID# 234015, Sankt Pölten, Lower Austria
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 228366, Salzburg, Salzburg
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 247510, Linz, Upper Austria
- Belgium (7):
  - Uza /Id# 228521, Edegem, Antwerpen
  - Hospital La Louviere Site Jolimont - Helora /ID# 228520, La Louvière, Hainaut
  - Groupe Sante CHC - Clinique du MontLegia /ID# 230415, Liège, Liege
  - Vitaz /Id# 228525, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 247780, Leuven, Vlaams-Brabant
  - Institut Jules Bordet /ID# 254676, Anderlecht
  - AZ Turnhout - Campus Sint-Elisabeth /ID# 231628, Turnhout
- Brazil (9):
  - Hospital de Clinicas da Universidade Federal do Parana /ID# 228123, Curitiba, Paraná
  - Instituto Nacional de Cancer (INCA) /ID# 228706, Rio de Janeiro, Rio de Janeiro
  - Upeclin Fmb - Unesp /Id# 252912, Botucatu, São Paulo
  - Hospital Amaral Carvalho - Fundacao Doutor Amaral Carvalho /ID# 228129, Jaú, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência /ID# 228121, São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino - Regional Sao Paulo /ID# 252918, São Paulo, São Paulo
  - Fundacao Antonio Prudente - AC Camargo Cancer Center /ID# 228130, São Paulo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual /ID# 230182, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 228127, São Paulo, São Paulo
- Canada (5):
  - Cross Cancer Institute /ID# 249080, Edmonton, Alberta
  - BC Cancer - Victoria /ID# 228850, Victoria, British Columbia
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 229896, Lévis, Quebec
  - CHUQ- Hôpital de l'Enfant-Jesus /ID# 231537, Québec, Quebec
  - CISSSBSL -Hopital regional de Rimouski /ID# 229894, Rimouski, Quebec
- China (24):
  - Peking University First Hospital /ID# 250517, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 230885, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 233919, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University /ID# 238427, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 231463, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital（Huifu Campus） /ID# 232512, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 230383, Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University /ID# 238657, Shijiazhuang, Hebei
  - Henan Cancer Hospital /ID# 230459, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 234153, Wuhan, Hubei
  - Hubei Cancer Hospital /ID# 232255, Wuhan, Hubei
  - Hunan Cancer Hospital /ID# 232153, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University /ID# 232511, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College /ID# 232513, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 231047, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital /ID# 232507, Nanchang, Jiangxi
  - The First Hospital of China Medical University /ID# 232509, Shenyang, Liaoning
  - Xijing Hospital /ID# 238650, Xi'an, Shaanxi
  - Fudan University Cancer Hospital /ID# 250475, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital /ID# 230876, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital /ID# 232062, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 230390, Hangzhou, Zhejiang
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 231250, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 231389, Hangzhou, Zhejiang
- Czechia (4):
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 228269, Hradec Králové, Hradec Kralove
  - Všeobecná Fakultní Nemocnice v Praze /ID# 228565, Prague, Praha 17
  - Fakultni nemocnice Kralovske Vinohrady /ID# 228564, Prague
  - Duplicate_Fakultni Nemocnice v Motole /ID# 228272, Prague
- Denmark (2):
  - Regionshospitalet Godstrup /ID# 227466, Herning, Central Jutland
  - Sygehus Lillebalt, Vejle /ID# 227404, Vejle, Region Syddanmark
- France (19):
  - CHU Clermont-Ferrand /ID# 238676, Clermont, Auvergne-Rhône-Alpes
  - CHU de Rennes - PONTCHAILLOU /ID# 230356, Rennes, Brittany Region
  - CHU Dijon /ID# 230354, Dijon, Cote-d Or
  - CHU Limoges - Dupuytren 1 /ID# 231450, Limoges, Franche-Comte
  - CHU NIMES - Hopital Caremeau /ID# 230351, Nîmes, Gard
  - Centre Hospitalier Universitaire de Bordeaux /ID# 230347, Pessac, Gironde
  - CHU Reims - Hôpital Robert Debre /ID# 248710, Reims, Marne
  - CHRU Nancy - Hopitaux de Brabois /ID# 241595, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 230353, Lille, Nord
  - IUCT Oncopole /ID# 233486, Toulouse, Occitanie
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 230358, Créteil, Paris
  - Hôpital Saint-Louis /ID# 232067, Paris, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 245928, Nantes, Pays de la Loire Region
  - Centre Leon Berard /ID# 230348, Lyon, Rhone
  - HCL - Hopital Lyon Sud /ID# 231449, Pierre-Bénite, Rhone
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 234095, La Roche-sur-Yon, Vendee
  - CHU Poitiers - La miletrie /ID# 230357, Poitiers, Vienne
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 245929, Caen
  - Hopital Pitie Salpetriere /ID# 230360, Paris, Île-de-France Region
- Germany (14):
  - Universitaetsklinikum Tuebingen /ID# 229663, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg /ID# 229278, Würzburg, Bavaria
  - Universitaetsklinikum Giessen /ID# 234245, Giessen, Hesse
  - Klinikum Kassel /ID# 229185, Kassel, Hesse
  - Universitaetsmedizin Goettingen /ID# 230411, Göttingen, Lower Saxony
  - Universitaetsklinikum Bonn /ID# 249401, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 229754, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 242907, Leipzig, Saxony
  - Otto-von-Guericke-Universitaet /ID# 230144, Magdeburg, Saxony-Anhalt
  - Helios Klinikum Berlin-Buch /ID# 229178, Berlin, State of Berlin
  - Universitaetsklinikum Jena /ID# 232064, Jena, Thuringia
  - Sozialstiftung Bamberg /ID# 229184, Bamberg
  - Universitaetsklinikum Essen /ID# 229180, Essen
  - Klinikum Mutterhaus der Borromäerinnen /ID# 232354, Trier
- Greece (7):
  - General Hospital of Athens Laiko /ID# 226626, Athens, Attica
  - Alexandra General Hospital /ID# 226632, Athens, Attica
  - University General Hospital Attikon /ID# 226629, Athens, Attica
  - University General Hospital of Ioannina /ID# 226628, Ioannina, Ioannina
  - General University Hospital of Thessaloniki AXEPA /ID# 226630, Thessaloniki, Thessaloniki
  - Theageneio Anticancer Hospital /ID# 226627, Thessaloniki, Thessaloniki
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 226633, Athens
- Hungary (8):
  - Semmelweis Egyetem /ID# 229291, Budapest, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 229286, Budapest, Budapest
  - Debreceni Egyetem-Klinikai Kozpont /ID# 229287, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 246475, Kaposvár, Somogy County
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 232203, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Szegedi Tudományegyetem /ID# 229289, Szeged, Szeged
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 229290, Szombathely, Vas County
  - Orszagos Onkologiai Intezet /ID# 229292, Budapest
- Israel (7):
  - Yitzhak Shamir Medical Center /ID# 228037, Ẕerifin, Central District
  - Rambam Health Care Campus /ID# 227849, Haifa, Haifa District
  - Hadassah /ID# 227846, Jerusalem, Jerusalem
  - ZIV Medical Center /ID# 232257, Safed, Northern District
  - The Chaim Sheba Medical Center /ID# 228322, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 228529, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 228043, Petah Tikva
- Italy (14):
  - Azienda Ospedaliero - Universitaria SS. Antonio e Biagio e Cesare Arrigo - Aless /ID# 227401, Alessandria, Alessandria
  - Duplicate_I.R.C.C.S Istituto Tumori Giovanni Paolo II /ID# 227400, Bari, Bari
  - ASST degli Spedali Civili di Brescia /ID# 227397, Brescia, Brescia
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 228458, San Giovanni Rotondo, Foggia
  - IRCCS Ospedale San Raffaele /ID# 228669, Milan, Milano
  - Istituto Europeo Di Oncologia /ID# 227396, Milan, Milano
  - Duplicate_Azienda Ospedaliera Universitaria Federico II /ID# 230403, Napoli, Napoli
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 227402, Palermo, Palermo
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 229820, Turin, Piedmont
  - Duplicate_Centro di Riferimento Oncologico /ID# 227395, Aviano, Pordenone
  - Ospedale Santa Maria Delle Croci /ID# 227394, Ravenna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 230402, Rome, Roma
  - Istituto di Candiolo Fondazione del Piemonte per l'Oncologia IRCCS /ID# 229602, Candiolo, Torino
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 227399, Novara
- Japan (24):
  - Duplicate_NHO Nagoya Medical Center /ID# 230678, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 230134, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 264541, Toyoake, Aichi-ken
  - National Cancer Center Hospital East /ID# 232423, Kashiwa-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 251866, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center /ID# 252245, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 230136, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 251839, Fukushima, Fukushima
  - Hokkaido University Hospital /ID# 231443, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 251945, Kobe, Hyōgo
  - Kagoshima University Hospital /ID# 232251, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 252135, Isehara, Kanagawa
  - Kitasato University Hospital /ID# 264668, Sagamihara-shi, Kanagawa
  - Kyoto University Hospital /ID# 231156, Kyoto, Kyoto
  - Mie University Hospital /ID# 251944, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 232303, Sendai, Miyagi
  - Shinshu University Hospital /ID# 252246, Matsumoto-shi, Nagano
  - Okayama University Hospital /ID# 232009, Okayama, Okayama-ken
  - Osaka City General Hospital /ID# 264670, Osaka, Osaka
  - Kindai University Hospital /ID# 232152, Osakasayama-shi, Osaka
  - National Cancer Center Hospital /ID# 230004, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 230271, Koto-ku, Tokyo
  - Yamagata University Hospital /ID# 230005, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital /ID# 263715, Kofu, Yamanashi
- Netherlands (12):
  - Canisius-Wilhelmina Ziekenhuis /ID# 248138, Nijmegen, Gelderland
  - Amphia Ziekenhuis /ID# 247739, Breda, North Brabant
  - Olvg /Id# 247899, Amsterdam, North Holland
  - Dijklander Ziekenhuis /ID# 248993, Hoorn, North Holland
  - Medisch Spectrum Twente /ID# 247854, Enschede, Overijssel
  - Universitair Medisch Centrum Groningen /ID# 247741, Groningen, Provincie Groningen
  - Albert Schweitzer Ziekenhuis /ID# 247740, Dordrecht, South Holland
  - Leids Universitair Medisch Centrum /ID# 247742, Leiden, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis /ID# 248139, Rotterdam, South Holland
  - St. Antonius Ziekenhuis /ID# 248644, Nieuwegein, Utrecht
  - Admiraal de Ruyter Ziekenhuis /ID# 247692, Goes, Zeeland
  - Deventer Ziekenhuis /ID# 247853, Deventer
- New Zealand (3):
  - Aotearoa Clinical Trials /ID# 228509, Papatoetoe, Auckland
  - North Shore Hospital /ID# 228508, Takapuna, Auckland
  - Palmerston North Hospital /ID# 232352, Palmerston North, Manawatu-Wanganui
- Poland (5):
  - ARS-MEDICAL Sp. z o.o. /ID# 229601, Piła, Greater Poland Voivodeship
  - Aidport Sp. z o.o. /ID# 229299, Skórzewo, Greater Poland Voivodeship
  - Pratia MCM Krakow /ID# 229121, Krakow, Lesser Poland Voivodeship
  - Szpitale Pomorskie Sp. z o.o /ID# 229122, Gdynia, Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej /ID# 229362, Kielce, Świętokrzyskie Voivodeship
- Puerto Rico (3):
  - Hematology and Oncology Institute /ID# 230056, Manatí, Puerto Rico
  - Pan American Center for Oncology Trials, LLC /ID# 230055, Rio Piedras, Puerto Rico
  - Auxilio Mutuo Cancer Center /ID# 248721, San Juan, Puerto Rico
- Narodny onkologicky ustav /ID# 239510, Bratislava, Bratislava Region, Slovakia
- South Africa (4):
  - Wits Clinical Research /ID# 228895, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 228896, Pretoria, Gauteng
  - University of Cape Town /ID# 228900, Cape Town, Western Cape
  - Haemalife Inc. /ID# 243392, Kuils River, Western Cape
- South Korea (10):
  - Inje University - Busan Paik Hospital /ID# 230293, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 228638, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 229798, Busan, Busan Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 228448, Seongnam-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 229800, Daegu, Gyeongsangbuk-do
  - Jeonbuk National University Hospital /ID# 228908, Jeonju, Jeonrabugdo
  - Seoul National University Hospital /ID# 228446, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 228444, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 228445, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 228447, Seoul, Seoul Teugbyeolsi
- Spain (15):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 228108, Badalona, Barcelona
  - Hospital Parc de Salut del Mar /ID# 228106, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 229859, Barcelona, Barcelona
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 228107, L'Hospitalet de Llobregat, Barcelona
  - Hospital San Pedro de Alcantara /ID# 248845, Cáceres, Caceres
  - Hospital Universitario Marques de Valdecilla /ID# 228984, Santander, Cantabria
  - Hospital Universitario Reina Sofia /ID# 228122, Córdoba, Cordoba
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 229157, Madrid, Madrid
  - MD Anderson Madrid /ID# 229860, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 228113, Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 228110, Madrid, Madrid
  - Hospital Universitario 12 de Octubre /ID# 228109, Madrid, Madrid
  - Clinica Universidad de Navarra - Pamplona /ID# 228116, Pamplona, Navarre
  - Hospital Universitario de Salamanca /ID# 228117, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio /ID# 228118, Seville, Sevilla
- Sweden (3):
  - Sunderby sjukhus /ID# 228165, Luleå, Norrbotten County
  - Sodra Alvsborgs sjukhus /ID# 228886, Borås, Västra Götaland County
  - Linkoping University Hospital /ID# 233520, Linköping, Östergötland County
- Switzerland (4):
  - Kantonsspital Aarau AG /ID# 229113, Aarau, Canton of Aargau
  - Kantonsspital St. Gallen /ID# 229117, Sankt Gallen, Canton of St. Gallen
  - EOC Ospedale Regionale di Bellinzona e Valli /ID# 228922, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden /ID# 253862, Chur, Kanton Graubünden
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 227384, Kaohsiung City, Kaohsiung
  - China Medical University Hospital /ID# 227379, Taichung, Taichung
  - Taichung Veterans General Hospital /ID# 227383, Taichung, Taichung
  - National Cheng Kung University Hospital /ID# 227381, Tainan, Tainan
- Turkey (Türkiye) (9):
  - Ankara Universitesi Fakultesi /ID# 227790, Ankara, Ankara
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 248202, Istanbul, Istanbul
  - Istanbul Florence Nightingale Hastanesi /ID# 229546, Istanbul, Istanbul
  - Duplicate_Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 227855, Istanbul, Istanbul
  - Ege University Medical Faculty /ID# 227792, Izmir, İzmir
  - Kocaeli University Med Faculty /ID# 227854, Köseköy, Kocaeli
  - Ondokuz mayis University Facul /ID# 227794, Samsun, Samsun
  - Akdeniz Universitesi Tip Fakul /ID# 227791, Antalya
  - Dicle Universitesi Tip /ID# 230087, Diyarbakır
- United Kingdom (11):
  - University Hospitals Birmingham NHS Foundation Trust /ID# 230043, Birmingham, Birmingham
  - Derriford Hospital and the Royal Eye Infirmary /ID# 230038, Plymouth, Devon
  - Gartnavel General Hospital /ID# 230027, Glasgow, Glasgow City
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 230028, London, Greater London
  - Clatterbridge Cancer Centre - Liverpool /ID# 230036, Liverpool, Liverpool
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 230123, Newcastle upon Tyne, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust /ID# 230035, Oxford, Oxfordshire
  - Leeds Teaching Hospitals NHS Trust /ID# 230471, Leeds, West Yorkshire
  - East Suffolk and North Essex NHS Foundation Trust /ID# 230040, Colchester
  - The Christie Hospital /ID# 230124, Manchester
  - Portsmouth Hospitals University NHS Trust /ID# 230044, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Falchi L, Nijland M, Huang H, Linton KM, Seymour JF, Tao R, Kwiatek M, Costa A, Vassilakopoulos TP, Greil R, Jimenez-Ubieto A, Gangatharan SA, Benjamini O, Thieblemont C, Tucci A, Elinder-Camburn A, Illes A, Novak J, Pavlovsky MA, McDonald A, Yoon DH, Maruyama D, Sunkersett G, Mei JP, Mukherjee N, Zhu F, Alshreef A, Favaro E, Morschhauser F; EPCORE FL-1 Investigators. Epcoritamab, lenalidomide, and rituximab versus lenalidomide and rituximab for relapsed or refractory follicular lymphoma (EPCORE FL-1): a global, open-label, randomised, phase 3 trial. Lancet. 2026 Jan 10;407(10524):161-173. doi: 10.1016/S0140-6736(25)02360-8. Epub 2025 Dec 7. PMID 41371238
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M20-638